CLINICAL TRIAL: NCT02236078
Title: Brief Bactericidal Activity of Anti-Tuberculosis Drugs in Drug-Resistant Tuberculosis
Brief Title: Brief Bactericidal Activity of Anti-Tuberculosis Drugs
Acronym: BBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHHSTP-6435
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-01

CONDITIONS: Tuberculosis; Drug-resistant Tuberculosis; Isoniazid Resistant Tuberculosis (Disorder)
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High dose isoniazid (Experimental): INH 900 mg daily to be administered orally for 6 days (600 mg for patients weighing <45 kg)
  Interventions: Drug: High dose isoniazid

INTERVENTIONS:
Drug: High dose isoniazid — See arm description
  Other Names: High dose INH

SUMMARY:
The investigators will determine the bactericidal activity of high-dose isoniazid against M. tuberculosis isolates that are (1) susceptible to isoniazid at 2.0 mcg/ml but resistant at 0.1 and 0.4 mcg/ml or (2) susceptible at 0.4 mcg/ml but resistant at 0.1 mcg/ml when tested in the BD MGIT 960 system. Further, the investigators will investigate the molecular genetic determinants of these differences in susceptibility.

To achieve these objectives the investigators will carry out an innovative variation on early bactericidal activity (EBA) study methodology. Patients at risk for drug-resistant TB will be screened for INH resistance using approved molecular assays. In those with INH-resistant TB, the investigators will quickly perform phenotypic DSTs using the direct method in the Bactec Mycobacterium Growth Indicator Tube (MGIT) 960 system, so results will be available within 7 days. If the DST results show the susceptibility patterns noted above, patients will receive 900 mg/d INH (600 mg if <45kg), and assess its effect with serial quantitative sputum cultures for 6 days. If the concentration of viable bacteria decreases significantly, the investigators will interpret this to mean the drug is having an effect. If not, the drug is ineffective. After 6 days, the patients will resume treatment according to national guidelines.

In case the investigators identify drugs that are effective under these conditions, the investigators will sequence known and putative genes associated with the action of these drugs for the mycobacterial isolates from these patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* INH resistance by approved molecular genetic test
* Phenotypic drug susceptibility test results match one of the required patterns
* Sputum microscopy positive for acid fast bacilli

Exclusion Criteria:

* Ineligible for MDR TB treatment according to national guidelines
* HIV infection with CD4 count less than 50
* Pregnancy
* Incarceration
* Too sick to participate (Karnofsky score <60, arterial pO2<90, respiratory rate repeatedly >25/min, clinician's judgment)
* Hepatic enzymes >3x normal
* Estimated glomerular filtration rate <60 mL/min/1.73 m2
* Unable to provide adequate sputum specimen

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Delta CFU/ml/day | 6 days
  Change in colony forming units per ml of sputum over 6 days

SECONDARY OUTCOMES:
Time-to-detection (TTD) | 6 days
  Interval in hours from culture inoculation to detection of mycobacterial growth in MGIT 960

OTHER OUTCOMES:
Acquired isoniazid resistance | 2 months
  Increased level of resistance to isoniazid

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E. Smith-Jeffcoat, MPH, Principal Investigator — U.S. Centers for Disease Control and Prevention; J. P. Cegielski, MD, MPH, Principal Investigator — JP Cegielski Consulting LLC
Locations (1):
- National Institute for Research on Tuberculosis, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Dalton T, Cegielski P, Akksilp S, Asencios L, Campos Caoili J, Cho SN, Erokhin VV, Ershova J, Gler MT, Kazennyy BY, Kim HJ, Kliiman K, Kurbatova E, Kvasnovsky C, Leimane V, van der Walt M, Via LE, Volchenkov GV, Yagui MA, Kang H; Global PETTS Investigators; Akksilp R, Sitti W, Wattanaamornkiet W, Andreevskaya SN, Chernousova LN, Demikhova OV, Larionova EE, Smirnova TG, Vasilieva IA, Vorobyeva AV, Barry CE 3rd, Cai Y, Shamputa IC, Bayona J, Contreras C, Bonilla C, Jave O, Brand J, Lancaster J, Odendaal R, Chen MP, Diem L, Metchock B, Tan K, Taylor A, Wolfgang M, Cho E, Eum SY, Kwak HK, Lee J, Lee J, Min S, Degtyareva I, Nemtsova ES, Khorosheva T, Kyryanova EV, Egos G, Perez MT, Tupasi T, Hwang SH, Kim CK, Kim SY, Lee HJ, Kuksa L, Norvaisha I, Skenders G, Sture I, Kummik T, Kuznetsova T, Somova T, Levina K, Pariona G, Yale G, Suarez C, Valencia E, Viiklepp P. Prevalence of and risk factors for resistance to second-line drugs in people with multidrug-resistant tuberculosis in eight countries: a prospective cohort study. Lancet. 2012 Oct 20;380(9851):1406-17. doi: 10.1016/S0140-6736(12)60734-X. Epub 2012 Aug 30. PMID 22938757